CLINICAL TRIAL: NCT02715713
Title: Autonomic Manifestations of Testosterone Deficiency in Men
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigator left the institution in August, 2016;
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Other Study IDs: L16-059
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Autonomic Neuropathy; Male Hypogonadism
Keywords: Autonomic neuropathy, Testosterone Deficiency
MeSH Terms: conditions — Eunuchism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- testosterone deficiency group: Men between the ages of 40 to 80-years-old with testosterone deficiency
- prostate cancer group: Men between the ages of 40 to 80-years-old with prostate cancer that will result in testosterone deficiency due to surgical or pharmacological castration.

SUMMARY:
The primary goal of this pilot study is to investigate the association between testosterone deficiency and the presence of abnormalities in the function of the autonomic nervous system. If such association exists, then we will investigate the effect of testosterone replacement therapy on correcting these abnormalities.

DETAILED DESCRIPTION:
The investigators will recruit 40 men between the ages of 40 to 80-years-old with low testosterone. Participants will be selected among those males referred to the Texas Tech University Health Sciences Center's (TTUHSC's) Internal Medicine Endocrinology Division outpatient clinic for the study and management of testosterone deficiency and to the TTUHSC Urology Department for diagnosis and management of prostate cancer that will result in testosterone deficiency due to surgical or pharmacological castration.

After recruitment, patients will have an initial standard clinical visit where aspects such as fatigue and anxiety will be investigated, followed by a full battery of autonomic testing (tilt table, heart rate response to deep breathing, Valsalva, and the Quantitative Sudomotor Axon Reflex Test (QSART).

Those patients with an initial diagnosis of testosterone deficiency will be initiated on testosterone replacement (intramuscular or skin routes) as standard of care, followed by a second visit in three (3) months--after normalization of serum testosterone levels--to evaluate changes in anxiety and fatigue level, and to repeat the cardiovascular autonomic function test.

Those patients with primary diagnosis of prostate cancer and normal serum testosterone levels will be evaluated a second time after confirmation of low testosterone, as described above. Standard questionnaires will be used to evaluate fatigue and anxiety. The autonomic testing of the heart will include tilt table (tilt the patient 70 degree by special designed table) and heart rate response to deep breathing, and Valsalva maneuver. Descriptive statistics will be compared between before and after treatment using different statistical methods.

ELIGIBILITY:
Inclusion Criteria for first group:

1. Patients with testosterone deficiency (total testosterone< 277 ng/dL [9.6 nmol/L]) measured between 7-10 am, and with one or more symptoms and signs suggestive of androgen deficiency as mainly determined by history.

   * Reduced sexual desire (libido)
   * Decreased spontaneous erections
   * Breast discomfort, gynecomastia
   * Loss of body (axillary and pubic) hair - reduced shaving
   * Very small (<5ml) or shrinking testes
   * Height loss
   * Low trauma fracture
   * Low bone mineral density
   * Hot flushes
   * Sweats
   * Decreased energy
   * Decreased motivation
   * Decreased initiative
   * Decreased self confidence
   * Feeling sad or blue
   * Depressed mood
   * Dysthymia
   * Poor concentration
   * Poor memory
   * Sleep disturbance
   * Increased sleepiness
2. Age 40 to 80 years

Inclusion Criteria for second group:

1. Patients who underwent chemical or surgical castration for prostatic cancer who are going to receive androgen deprivation therapy.
2. Age 40 to 80 years

Exclusion Criteria (both groups):

1. Patients with history or current diagnosis of:

* Atrial fibrillation.
* Cardiac arrythmia
* Pacemaker placement.
* Myocardial infarction < 3 months
* Uncontrolled diabetes mellitus with hemoglobin A1c > 8.5% in the last 6 months.
* Diabetes mellitus with autonomic neuropathy
* Breast cancer
* Heart failure with left ventricular ejection fraction below 35%.
* Severe sleep apnea.
* Recent eye surgery (< 3 months)
* Recent ischemic stroke (< 3 months)
* History of retinal detachment.
* History of brain aneurysm.
* Severe chronic obstructive pulmonary disease (COPD) on oxygen therapy.
* Intraocular hemorrhage and lens dislocation.
* Glaucoma.
* Thyroid disease.
* Not literate in English

Exclusion Criteria for patient who will receive testosterone treatment

* Metastatic prostate cancer
* Prostate-specific antigen (PSA) concentration >4.0 mcg/L,
* Prostate-specific antigen (PSA) >3.0 mcg/L in high-risk men (African-Americans or men with first-degree relatives with prostate cancer). (Measured at clinic visit 1)
* Polycythemia (hemoglobin level >18 g/dL, hematocrit > 52%) (measured at clinic visit 1)
* Severe acne.
* History of venous or arterial thrombosis.
* Persons not literate in English

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two groups will be recruited with 20 men in each group:
  Group 1 will include 20 men between the ages of 40 to 80-years-old with symptoms and biochemical parameters of low testosterone.
  Group 2 will include 20 men between the ages of 40 to 80-years-old with prostate cancer and normal serum testosterone that will be treated with surgical or pharmacological castration, as following standard of care at Urology Division, resulting in testosterone deficiency.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with testosterone deficiency who will have abnormal autonomic function test (abnormal heart rate response to deep breathing, abnormal Valsalva ratio, and abnormal tilt table i.e. orthostatic hypotension). | 24 months

SECONDARY OUTCOMES:
Number of patients with testosterone deficiency and abnormal autonomic function test who will have such abnormalities corrected if they receive testosterone replacement therapy as part of standard of care. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Eldokla, MD, Principal Investigator — Texas Tech Universty Health Science Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided